CLINICAL TRIAL: NCT07095933
Title: The Safety and Efficacy Evaluation of Everolimus as an Adjunctive Treatment for Focal Refractory Epilepsy: A Pilot Study
Brief Title: The Safety and Efficacy Evaluation of Everolimus as an Adjunctive Treatment for Focal Refractory Epilepsy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-218-002
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Drug Resistant
Keywords: Everolimus; Focal Refractory Epilepsy; Epilepsy memory; mTOR pathway
MeSH Terms: conditions — Epilepsy | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): All subjects will receive the experimental drug.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Oral administration is given solely for the epilepsy seizure event. Dosage: The dosage is determined based on body surface area (BSA), with 2.5 mg per dose for BSA <1.2 m², 5 mg per dose for BSA 1.3-2.1 m², and 7.5 mg per dose for BSA >2.2 m².

SUMMARY:
The aim of this study is to evaluate the clinical efficacy of everolimus as an adjunctive therapy for refractory epilepsy. The significance lies in addressing whether the mTOR inhibitor sirolimus has antiepileptic adjunctive effects for a broader range of patients with refractory epilepsy, with the hope of providing a new mTOR-targeted antiepileptic adjunctive medication regimen that is administered only during epileptic events and can be widely used for various types of refractory epilepsy.

DETAILED DESCRIPTION:
Previous research has shown that the mTOR pathway is involved in the "epilepsy memory" process. Associating the acute seizures of the mouse kainic acid epilepsy model with a specific odor stimulus can lead to specific induction of epileptic seizures by this odor stimulus two weeks later. After epileptic seizures induced by a specific odor stimulus, the expression of the memory-related molecule pmTOR in the mouse hippocampus changes in a time-dependent manner, indicating that the mTOR signaling pathway is involved in the reconsolidation process of epilepsy memory. Further intervention in the reconsolidation process of epilepsy memory with the mTOR inhibitor everolimus (Rap) found that administering the drug within the memory consolidation window (5 min) could effectively intervene in the reinduction of epilepsy, while administering the drug outside the memory consolidation window (9 h) could not intervene. Professor Huang Zhuo's team validated the above experimental results using a conditioned epilepsy memory mouse model. Clinical experiments have found that administering the mTOR pathway inhibitor everolimus immediately after an epileptic seizure in patients can significantly reduce the interictal brain electrical activity, showing promising epilepsy treatment effects. However, this study only involved a single drug treatment, the treatment duration was short, and only the changes in epileptiform discharges after treatment with everolimus in epileptic patients were evaluated at the electrophysiological level, without evaluating the control efficacy on seizure symptoms in patients after repeated seizures with a sufficient course of treatment.

Therefore, inhibiting the mTOR signaling pathway within a specific time window by intervening in the reconsolidation of the current epileptic event holds promise as a new strategy to alleviate subsequent seizures. This strategy is expected to be applicable to a broader range of treatments for refractory epilepsy, and administering medication only during epileptic events is anticipated to achieve more efficient therapeutic effects.

Everolimus (sirolimus) is an inhibitor of the mammalian target of rapamycin (mTOR). In studies using animal models of tuberous sclerosis complex (TSC), mTOR inhibitors have been found to significantly reduce the frequency of epileptic seizures; furthermore, everolimus is currently undergoing phase III clinical trials as an adjunctive treatment for refractory epilepsy associated with TSC. Evidence from various animal models of epilepsy, including genetic epilepsy (such as in WAG/Rij rats) and acquired epilepsy (such as those induced by kainic acid or pilocarpine), also suggests the involvement of the mTOR signaling pathway in these forms of epilepsy and the broad inhibitory effects of mTOR inhibitors on epileptic seizures.

Based on the "epilepsy memory" mechanism, combining everolimus with a memory reconsolidation paradigm holds promise as an effective adjunctive treatment for refractory epilepsy. Evaluating its efficacy and safety not only helps establish its value in epilepsy treatment but also provides important guidance for clinical practice, crucial for the transition from basic research to clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years (inclusive), regardless of sex.
* Diagnosis of epilepsy, meeting the criteria for focal seizures or focal to bilateral tonic-clonic seizures as defined by the 2017 International League Against Epilepsy (ILAE) classification.
* History of epileptic seizures lasting ≥30 seconds, accompanied by impaired awareness.
* At least 16 focal seizures during the 8-week baseline period prior to enrollment, with no seizure-free interval of 21 consecutive days.
* Findings on electroencephalography (EEG) or neuroimaging (MRI or CT) performed within 2 years prior to screening consistent with a diagnosis of focal epilepsy, and exclusion of progressive structural central nervous system lesions or progressive encephalopathy.
* Diagnosis of drug-resistant epilepsy, defined as failure to achieve sustained seizure freedom despite adequate trials of at least two appropriately chosen and tolerated antiseizure medications (ASMs) over a period of 2 years. - Existing ASMs must have no known drug-drug interactions with everolimus and must have been administered at a stable dose for at least 12 weeks prior to enrollment.
* Use of vagus nerve stimulation (VNS) or deep brain stimulation (DBS) is permitted, provided the device was implanted at least 5 months prior to screening, with stimulation parameters stable for at least 12 weeks before enrollment and maintained unchanged throughout the study.
* Written informed consent to participate in the study, provided voluntarily by the subject.
* In the investigator's judgment, the subject is able to comply with the requirements of the study protocol, including understanding and completing seizure diaries, adhering to the visit schedule, and taking study medications as directed.

Exclusion Criteria:

* Diagnosis of primary generalized epilepsy.
* History of non-epileptic events (e.g., psychogenic non-epileptic seizures).
* Patients with only non-motor focal seizures according to the 2017 ILAE classification.
* Epilepsy with identifiable and treatable causes (e.g., metabolic disorders, intoxication, infection, space-occupying lesions, or confirmed genetic abnormalities).
* Inability to accurately count seizures due to excessively frequent episodes within the 12 months prior to study drug administration.
* History of epileptic seizure clusters within the 12 months prior to study drug administration.
* History of status epilepticus within the 12 months prior to study drug administration.
* Use of mTOR pathway inhibitors within the 12 months prior to study drug administration.
* History of cerebrovascular events (e.g., cerebral infarction, cerebral hemorrhage, or transient ischemic attack) or progressive intracranial lesions within the 6 months prior to study drug administration.
* Presence of severe uncontrolled diseases, including immunodeficiency disorders, hepatic or renal disease, acute infection, significant pulmonary dysfunction, or advanced malignancy.
* Severe cardiovascular or peripheral vascular disease, such as New York - Heart Association (NYHA) class III-IV heart failure, malignant arrhythmias (e.g., long QT syndrome, Brugada syndrome, conduction block), any other clinically significant ECG abnormalities, or myocardial infarction within 3 months prior to screening.
* History of any condition or surgery that, in the investigator's opinion, could affect absorption, distribution, or metabolism of the study drug (e.g., active gastric ulcer, ulcerative colitis, Crohn's disease, intestinal obstruction), or presence of dysphagia.
* Any medical condition, psychiatric disorder, cognitive impairment, or intellectual disability that, in the investigator's judgment, may increase the risk to the subject or interfere with study participation.
* Laboratory abnormalities meeting any of the following criteria: alanine aminotransferase (ALT) >2× upper limit of normal (ULN), aspartate aminotransferase (AST) >2× ULN, alkaline phosphatase (ALP) >2× ULN, platelet count <80×10⁹/L, neutrophil count <1.8×10⁹/L, or creatinine clearance (CLcr) <30 mL/min (calculated by the Cockcroft-Gault formula).
* Female subjects who test positive for pregnancy during screening or who are breastfeeding.
* History of alcohol or substance abuse within 2 years prior to study drug administration.
* Participation in any other clinical trial within 3 months prior to study drug administration, except for non-interventional clinical trials.
* Known hypersensitivity or allergy to any component of everolimus tablets.
* Current use of medications that may affect the central nervous system or the metabolism of everolimus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Seizure Frequency Per 28 Days | assessed per 28 days during the treatment until the end of 12-week treatment.
  Percent change in 28-day frequency of seizures during the 12 week treatment and follow-up period relative to baseline

SECONDARY OUTCOMES:
50% Seizure Responder Rate | Baseline observation period, and 12-week treatment period (ending at 12 weeks).
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Seizure Severity | Baseline observation period, and 12-week treatment period (ending at 12 weeks).
  The percent change from baseline in seizure severity evaluated by Liverpool seizure severity scale (LSSS) .
Life quality evaluation | Baseline observation period, and 12-week treatment period (ending at 12 weeks).
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Adverse Events | through study completion, 12 weeks.
  Rate of adverse events which were judged to be study-related throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No